CLINICAL TRIAL: NCT05766696
Title: Survival Rate and Cost-effectiveness of Glass Ionomer Restorations in the Primary Molars Using ART and Conventional Cavity Preparations in South African Children: a Randomized Controlled Non Inferiority Trial
Brief Title: Survival Rate and Cost-effectiveness of Conventional vs ART Restorations in a School Setting
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: DMG Dental Material Gesellschaft mbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: DeltaART
Record Dates: First submitted 2023-03-02; First posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Dental Caries
Keywords: Glass Ionomer Cements; Atraumatic Restorative Treatment; Cost Effectiveness; Oral Health
MeSH Terms: conditions — Dental Caries | interventions — Dental Atraumatic Restorative Treatment

STUDY DESIGN:
Intervention Model Description: This study is a parallel-group, randomized, controlled non-inferiority trial with a 2-year follow up. School children (from 2 schools) in a township in South Africa are randomized to the ART group (class room) or Conventional group (mobile clinic).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atraumatic Restorative Treatment (ART) (Experimental): GIC restorations placed using ART in a class room.
  Interventions: Procedure: Atraumatic Restorative Treatment (ART)
- Conventional Cavity Preparation (Active Comparator): GIC restorations placed using conventional cavity preparation in a mobile clinic.
  Interventions: Procedure: Conventional Cavity Preparation

INTERVENTIONS:
Procedure: Atraumatic Restorative Treatment (ART) — Conventional glass-ionomer restorations are placed using the Atraumatic Restorative Treatment (ART) technique. Essentially, cavities are prepared using hand instrument excavators. Afterwards, the cavity is conditioned (using a 10% polyacrylic acid conditioner) and cleaned, with subsequent insertion of a conventional restorative glass-ionomer. During the curing phase, Vaseline will be applied to all restoration surfaces for moisture protection.
  The treatment will be conducted in a class room.
  As concomitant treatment, all participants will receive supervised toothbrushing during the study using 1,450 ppm fluoride toothpaste once a day.
  Arms: Atraumatic Restorative Treatment (ART)
Procedure: Conventional Cavity Preparation — Conventional glass-ionomer restorations are placed after conventional cavity preparation. Essentially, cavities are prepared using rotary instruments/diamond burs. Afterwards, the cavity is conditioned (using a 10% polyacrylic acid conditioner) and cleaned, with subsequent insertion of a conventional restorative glass-ionomer. During the curing phase, Vaseline will be applied to all restoration surfaces for moisture protection.
  The treatment will be conducted in a mobile clinic.
  As concomitant treatment, all participants will receive supervised toothbrushing during the study using 1,450 ppm fluoride toothpaste once a day.
  Arms: Conventional Cavity Preparation

SUMMARY:
This study will investigate the performance and cost-effectiveness of glass-ionomer restorations placed in school children in an outreach setting in rural areas in South Africa over a 2-year period, when placed using either ART (in a classroom) or conventional (in a mobile clinic) cavity preparation.

DETAILED DESCRIPTION:
Access to dental care in South African townships is very limited, as indicated by a caries prevalence of 84% and severity of 4.9 (dmft) in 6 year olds. To tackle this burden school-based tooth-brushing programs have been suggested to be cost-effective while reducing inequalities in accessibility. However, despite their efforts, the caries burden remains high.

Alternatives are mobile dental services or treatment techniques that do not require extensive equipment such as Atraumatic Restorative Treatment (ART). Mobile dental services are more cost-effective than stationary clinics, but the costs of acquiring, outfitting, and running a mobile dental truck are factors that may hamper the broader use of this model. ART on the other hand is easy to execute with minimal equipment and monetary resources. But the drawback is a typically lower survival rate of ART restorations compared to conventional placed restorations.

This study aims to further assess and compare the performance and cost-effectiveness of glass-ionomer restorations when placed using either ART (in a classroom) or conventional (in a mobile clinic) cavity preparation in South African school children stemming from a periurban area. The results of this research may help to assess and implement future oral health care programs.

ELIGIBILITY:
General Inclusion Criteria:

* Children (4-8 years of age)
* Guardians have given informed consent
* Child is cooperative and assented

Inclusion criteria for teeth

* Cavity > 1 mm
* Tooth has no pathological mobility
* Tooth has no preexisting developmental defects
* Tooth has no pulp exposure or is indication for endodontic treatment
* No pain, fistula or abscess related to the selected tooth

Exclusion criteria for teeth

* Cavity > 1 mm
* Tooth has no pathological mobility

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Survival rate of posterior occlusal multi-surface restorations | 24 months
  Restorations are assessed using the ART criteria by Frencken:
  Survival: Code 0 (Present, satisfactory); Code 1 (Present, slight deficiency at cavity margin of less than 0.5 mm)
  Failure: Code 2 (Present, deficiency at cavity margin of 0.5 mm or more); Code 3 (Present, fracture in restoration); Code 4 (Present, fracture in tooth); Code 5 (Present, overextension of approximal margin of 0.5 mm or more); Code 6 (Not present, most or all of restoration missing); Code 7 (Not present, other restorative treatment performed); Code C (Dentin carious lesion present)

SECONDARY OUTCOMES:
Survival rate of restorations depending on lesion type (occlusal single surface, occlusal multi surface and approximal restorations) | 6, 12 and 24 months
  Restorations are divided in the subgroups "occlusal single surface", "occlusal multi surface" and "approximal restorations" and restorations are assessed using the ART criteria by Frencken:
  Survival: Code 0 (Present, satisfactory); Code 1 (Present, slight deficiency at cavity margin of less than 0.5 mm)
  Failure: Code 2 (Present, deficiency at cavity margin of 0.5 mm or more); Code 3 (Present, fracture in restoration); Code 4 (Present, fracture in tooth); Code 5 (Present, overextension of approximal margin of 0.5 mm or more); Code 6 (Not present, most or all of restoration missing); Code 7 (Not present, other restorative treatment performed); Code C (Dentin carious lesion present)
Incremental cost-effectiveness ratio (ICER) | 6, 12 and 24 months
  Incremental cost-effectiveness ratio will be calculated as "difference in costs of failures / difference in failures" to assess "cost/ savings per failure prevented".
  For costing, a payers perspective will be assumed and costing will be calculated on a "per restoration" basis. For this material, transport, personnel and equippment costs will be assessed. All materials used in each procedure will have their specifications and quantity registered. Capital costs will be annualized and the proportion of time it took to complete the intervention will be calculated and applied to the annualized capital costs to estimate the cost per restoration. Prices will be inferences from the market value converted in US Dollars and obtained by the medium of the values from different places that commercialized the referred products.

OTHER OUTCOMES:
Lesion size | Intervention at baseline
  Lesion size (<3.5mm; 3.5mm-5.5mm; >5.5mm) will be recorded to evaluate the impact of lesion size on survival rate
Treatment time (continuous outcome, minutes) | Intervention at baseline
  Treatment time (from lifting intrument to placing instrument) for each restoration will be recorded using a stopwatch

CONTACTS AND LOCATIONS:
Locations (1):
- Nyameko and Itsitsa Primary Schools, Mfuleni, Western Cape, South Africa